CLINICAL TRIAL: NCT02292017
Title: A Prospective Single Center Trial Investigating the Effects of Prospectively Measuring Packing Density Prior to Choosing Target Coils for the Treatment of Intracranial Saccular Aneurysms.
Brief Title: Prospective Packing Density With Target Coils I
Acronym: PropackI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Tennessee Neurovascular Institute, LLC (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TNVI 001
Record Dates: First submitted 2014-11-12; First posted 2014-11-17 (Estimated); Last update posted 2018-09-11 (Actual); Status verified 2018-09

CONDITIONS: Intracranial Aneurysm
MeSH Terms: conditions — Intracranial Aneurysm

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Embolization of intracranial aneurysm (Experimental): Embolization with Target Coils
  Interventions: Device: Embolization of intracranial aneurysm

INTERVENTIONS:
Device: Embolization of intracranial aneurysm — Cerebral angiogram will be performed, target aneurysm measurements are performed including dome height, width, and depth as well as the neck length. Aneurysm volume will be calculated. During the embolization, framing, filling, and finishing should be done with Target Coils. In the event of aneurysms with a wide neck a Neuroform Stent may be used to ensure the best clinical and angiographic outcome. Immediate post procedure angiography is performed using the same pre-treatment views to assess results and complications.
  Other Names: Coiling procedure

SUMMARY:
This is a prospective single center trial investigating the effects of prospectively measuring packing density prior to choosing Target Coils for the treatment of intracranial saccular aneurysms. Up to 25 eligible subjects with ruptured or unruptured intracranial saccular aneurysms between 4-20mm (maximum dimension), who consent to study participation, will be treated with Stryker Target Detachable Coils.

Historical data from patients enrolled in the MAPS trial at the single center will be the control arm of the trial and reviewed for comparison to the prospective arm. In the control arm, the subjects received Stryker Matrix2 Detachable Coils and Guglielmi Detachable Coils and packing density was not measured prior to these procedures. The Pro-Pack Trial will evaluate the outcomes of the subjects treated with Target Coils, in whom the packing density will be actively calculated prior to coil selection. This will serve to establish that a higher packing density can be obtained by the change in methodology of coil selection and a higher packing density with lower recurrence rates.

DETAILED DESCRIPTION:
The Pro Pack Trial will evaluate the outcomes of subjects treated with Target Coils, in whom the packing density is actively calculated prior to coil selection. Selecting the coil with the best volumetric filling has been shown to increase overall packing density. Each coil thereafter will be evaluated prior to placement to assess the resultant packing density. An initial goal of 10% or greater packing density with the first coil will be used as a guide to coil selection. A final packing density of greater than 25% should be attempted as feasible. Currently, a maximum packing density is not defined. While theoretically a packing density may approach 100%, in reality the spaces between the coil loops occupy a large percentage of the coil mass, and packing densities rarely reach 50% or greater. As such, the final packing density is left to the operator, and is based on ability to place coils safely by the operator.

Potential subjects will be screened, consented, imaged, and evaluated in order to obtain 25 patients with complete 12-month follow-up. Baseline patient data will be collected at the time of the procedure; follow-up information will be collected within 48 hours of the procedure, and at approximately 12 months (±3 months) after the procedure. The anticipated study duration is approximately 24 months: 12 month recruitment, 12 month primary endpoint and closeout.

Enrollment in the study occurs after a signed Informed Consent form has been obtained, all eligibility criteria have been met, aneurysm volume has been calculated, and the procedure to place Target Coils with prospective density measurements has begun, i.e., at the time of target procedural angiography. From the moment of placement of the first coil, the patient is considered in the study whether they receive Target Coils or not, and will be followed up and included in the final analysis. Patients enrolled in the trial will be followed for approximately 12 months after the index embolization procedure. This will allow evaluation of the primary and secondary study endpoints. Targeted enrollment is 25 patients with complete 12 month follow-up evaluations. Every effort will be made to follow the progress and monitor the safety of patients who have been treated with Target® Coils.

Embolization utilizing Target® Coils may proceed at the time of diagnostic angiography for eligible patients who have signed an Informed Consent form. The investigator must perform the embolization procedure. Framing, filling, and finishing should be done with Target Coils. In the event of aneurysms with wide necks or unfavorable anatomy, adjunctive therapy, Neuroform Stent may be used to ensure the best clinical and angiographic results.

The site will enter ongoing, real time information into an electronic imaging database and track outcomes during the follow-up angiographic evaluations. The degree of occlusion, by coils and/or thrombus, will be measured post procedurally and at 12 +/- 3 months post procedure by the Angiographic Core Laboratory using a 3 point categorical scale: complete, residual neck/dog ear or residual aneurysm. Additionally, for the final angiogram, a same/ better / worse scale shall be applied.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is between 18 and 85 years of age (inclusive).
2. Patient has a documented untreated intracranial saccular aneurysm 4-20 mm diameter angiographic lumen, ruptured or unruptured, suitable for embolization with coils.
3. Target® Coils are considered a treatment option. Every attempt should be made to treat with Target coils as possible to achieve optimal occlusion.
4. Target aneurysm can be adequately coiled at index procedure (NO staged coiling procedures).
5. Target aneurysm morphology allows for adequate retention of coils within the aneurysmal sac without occlusion of the parent artery, as determined by the treating physician.
6. Patient or patient's legally authorized representative has provided written informed consent.
7. Patient is willing and able to comply with protocol follow-up requirements.

Exclusion Criteria:

Candidates must be excluded from the study if ANY of the following criteria are met at the time of screening:

1. Patient is <18 or >80 years old.
2. Target aneurysm is not saccular in nature (mycotic, fusiform, and dissecting).
3. Target aneurysm is >20 mm maximum luminal dimension, <4 mm maximum luminal dimension.
4. Target aneurysm has been previously treated by surgery or endovascular therapy.
5. Target aneurysm is in the physician's estimation unlikely to be successfully treated by endovascular techniques.
6. Patient presents as Hunt and Hess grade IV or V for a ruptured aneurysm.
7. Patient presents with Modified Rankin Score 4 or 5 at baseline.
8. Patient is concurrently enrolled in another investigational drug or device study unless the sponsor grants permission.
9. Patient has known hypersensitivity to platinum, nickel, stainless steel or structurally related compounds found in Target® Coils.
10. Patients who have had or could have a severe reaction to contrast agents that cannot be adequately pre-medicated prior to the coiling procedure.
11. Patients who are unable to complete scheduled follow up assessments at the enrolling center due to limited life expectancy (<12 months), comorbidities or geographical considerations.
12. Planned use of adjunctive therapy stents except Neuroform is not allowed.
13. Patients with Moya-Moya disease, AVMs, arteriovenous fistula, intracranial tumors, intracranial hematoma (unrelated to target aneurysm), significant atherosclerotic stenosis, tortuosity or other conditions preventing access to the target aneurysm.

15. Target aneurysm with significant thrombosis that may increase the likelihood of recanalization at the discretion on the investigator.

16. Female patient has a positive pregnancy assessment at baseline.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2014-10; Primary Completion 2018-02-01 (Actual); Study Completion 2019-08-01 (Estimated)

PRIMARY OUTCOMES:
Packing density | 24 hours
  Increased packing density defined as an relative increase by 20% compared to the control arm after initial treatment.

SECONDARY OUTCOMES:
Target Aneurysm Recurrence (TAR) | Up to 15 months
  Angiographic assessments performed at 12-15 months consisting of residual aneurysm (Modified Raymond Scale) Complete, residual neck, or residual aneurysm.
Change of aneurysm filling | 12-15 months
  Same Better Worse Scale: The percentage of patients who experience any increase/decrease or no change of the aneurysm filling compared to initial post-treatment angiogram.
Technical Procedure Success | 24 hours
  Successful delivery and deployment of Target coils in the target aneurysm without intraoperative rupture.
Neurological morbidity/mortality | 12-15 months
  Measure functional outcomes by modified Rankin Scale

CONTACTS AND LOCATIONS:
Overall Officials: Keith Woodward, MD, Principal Investigator — Tennessee Neurovascular Institute, LLC
Locations (1):
- Fort Sanders Regional Medical Center, Knoxville, Tennessee, United States